CLINICAL TRIAL: NCT03038880
Title: STAIRWAY: Simultaneous Blockade of Angiopoietin-2 and VEGF-A With the Bispecific Antibody RO6867461 (RG7716) for Extended Durability in the Treatment of Neovascular Age-Related Macular Degeneration
Brief Title: Study to Evaluate Faricimab (RO6867461; RG7716) for Extended Durability in the Treatment of Neovascular Age Related Macular Degeneration
Acronym: STAIRWAY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR39521
Record Dates: First submitted 2017-01-31; First posted 2017-02-01 (Estimated); Results first posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Neovascularization, Choroidal; Macular Degeneration, Age-Related
MeSH Terms: conditions — Choroidal Neovascularization; Macular Degeneration | interventions — faricimab; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 6 mg Faricimab Q12W (Experimental): 6 mg faricimab was given by intravitreal (IVT) injection once every 4 weeks (Q4W) up to Week 12 (4 injections), followed by 6 mg faricimab IVT injection once every 12 weeks (Q12W) from Week 24 up to Week 48 (injections at Weeks 24, 36, and 48; 3 injections).
  Interventions: Drug: Faricimab; Drug: Sham Procedure
- 6 mg Faricimab Q16W (Experimental): 6 mg faricimab was administered by IVT injection once every 4 weeks (Q4W) up to Week 12 (4 injections), followed by no doses up to Week 24 when a protocol-defined assessment of disease activity was performed. Participants with disease activity at Week 24 initiated 6 mg faricimab IVT Q12W dosing, and participants without disease activity at Week 24 initiated 6 mg faricimab IVT once every 16 weeks (Q16W) dosing for the remainder of the study.
  Interventions: Drug: Faricimab; Drug: Sham Procedure
- 0.5 mg Ranibizumab Q4W (Active Comparator): 0.5 mg of ranibizumab was administered by IVT injection once every 4 weeks (Q4W) for 48 weeks (13 injections).
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Faricimab — Faricimab was administered via IVT injections as specified during the treatment period.
  Other Names: RO6867461; RG7716
  Arms: 6 mg Faricimab Q12W; 6 mg Faricimab Q16W
Drug: Ranibizumab — Ranibizumab was administered via IVT injections as specified during the treatment period.
  Other Names: Lucentis®
  Arms: 0.5 mg Ranibizumab Q4W
Drug: Sham Procedure — The sham was a procedure that mimicked an IVT injection and involved the blunt end of an empty syringe (without a needle) being pressed against the anesthetized eye. It was administered to participants in the faricimab treatments arms at applicable visits to maintain masking among treatment arms.
  Arms: 6 mg Faricimab Q12W; 6 mg Faricimab Q16W

SUMMARY:
This was a Phase II, multicenter, randomized, active comparator-controlled, 52-week study to investigate the efficacy, safety and pharmacokinetics of faricimab (RO6867461; RG7716) administered with extended dosing regimens in treatment-naive participants with neovascular age related macular degeneration (nAMD). Only one eye was chosen as the study eye.

ELIGIBILITY:
Inclusion Criteria

* Treatment-naive CNV secondary to AMD (nAMD)
* Subfoveal or juxtafoveal CNV with a subfoveal component related to the CNV activity by fundus fluorescein angiography (FFA) or spectral-domain optical coherence tomography (SD-OCT; as evidenced by subretinal fluid, subretinal hyperreflective material, evidence of leakage, or hemorrhage)
* CNV lesion of all types with: total lesion size (including blood, atrophy, fibrosis, and neovascularization) of 6 disc areas or less by FFA; and CNV component area of at least 50% of total lesion size by FFA; and active CNV confirmed by FFA (evidence of leakage); and CNV exudation confirmed by SD-OCT (presence of fluid)
* BCVA letter score of 73 to 24 letters (inclusive) on ETDRS-like charts (20/40-20/320 Snellen equivalent) on day 1
* Clear ocular media and adequate pupillary dilatation to allow acquisition of good-quality retinal images to confirm diagnosis

Exclusion Criteria:

* CNV due to causes other than AMD, such as ocular histoplasmosis, trauma, pathological myopia, angioid streaks, choroidal rupture, or uveitis
* Central serous chorioretinopathy at screening
* Retinal pigment epithelial tear involving the macula
* On FFA: subretinal hemorrhage, fibrosis, or atrophy of more than (>)50% of the total lesion area and/or that involves the fovea
* Any prior or concomitant treatment for CNV including (but not restricted to) IVT treatment (steroids, anti-VEGF, tissue plasminogen activator, ocriplasmin, C3F8 gas, air), periocular pharmacological intervention, argon laser photocoagulation, verteporfin photodynamic therapy, diode laser, transpupillary thermotherapy, or surgical intervention
* Cataract surgery within 3 months of baseline assessments
* Any other intraocular surgery (pars plana vitrectomy, glaucoma surgery, corneal transplant, radiotherapy)
* Prior IVT treatment (including anti-VEGF medication) except for management of cataract complication with steroid IVT treatment
* Prior periocular pharmacological intervention for other retinal diseases
* Any concurrent intraocular condition in the study eye (eg, amblyopia, aphakia, retinal detachment, cataract, diabetic retinopathy or maculopathy, or epiretinal membrane with traction) that, in the opinion of the investigator, could either reduce the potential for visual improvement or require medical or surgical intervention during the course of the study
* Active intraocular inflammation (grade trace or above) in the study eye on day 1 (before randomization)
* Current vitreous hemorrhage in the study eye
* Uncontrolled glaucoma (eg, progressive loss of visual fields or defined as IOP ≥25 mm Hg despite treatment with antiglaucoma medication) in the study eye
* Spherical equivalent of refractive error demonstrating more than 8 diopters of myopia in the study eye
* History of idiopathic or autoimmune-associated uveitis in either eye
* Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye on day 1 (before randomization)
* Any major illness or major surgical procedure within 1 month before screening
* Uncontrolled blood pressure (defined as systolic >180 mm Hg and/or diastolic >100 mm Hg while participant at rest). If a participant's initial reading exceeded these values, a second reading was taken later on the same day, or on another day during the screening period. If the participant's blood pressure was controlled by antihypertensive medication, the participant was taking the same medication continuously for at least 30 days before day 1
* Stroke or myocardial infarction within 3 months before day 1
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory findings giving reasonable suspicion of a condition that contraindicated the use of the investigational drug or that might affect interpretation of the results of the study or renders the participant at high risk for treatment complications in the opinion of the investigator
* Pregnant or breastfeeding, or intended to become pregnant during the study
* Known hypersensitivity to ranibizumab, fluorescein, any ingredients of the formulation used, dilating eye drops, or any of the anesthetic and antimicrobial drops used
* Treatment with investigational therapy within 3 months before initiation of study treatment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2017-01-27 (Actual); Primary Completion 2018-01-11 (Actual); Study Completion 2018-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (25):
- United States (25):
  - Retinal Consultants of Arizona, Phoenix, Arizona
  - Retina Associates Southwest PC, Tucson, Arizona
  - California Retina Consultants, Bakersfield, California
  - Retinal Diagnostic Center, Campbell, California
  - Retina Consultants of Southern Colorado PC; Clinical Research Department, Colorado Springs, Colorado
  - Rand Eye, Deerfield Beach, Florida
  - Florida Eye Associates, Melbourne, Florida
  - Retina Vitreous Assoc of FL, St. Petersburg, Florida
  - Southern Vitreoretinal Assoc, Tallahassee, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Midwest Eye Institute, Indianapolis, Indiana
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - The Retina Care Center, Baltimore, Maryland
  - Vitreo Retinal Surgery, Minneapolis, Minnesota
  - Sierra Eye Associates, Reno, Nevada
  - Eye Associates of New Mexico, Albuquerque, New Mexico
  - Vitreoretinal Consultants, Great Neck, New York
  - Oregon Retina, LLP, Eugene, Oregon
  - Retina Northwest, Portland, Oregon
  - Charles Retina Institute, Germantown, Tennessee
  - Retina Res Institute of Texas, Abilene, Texas
  - Texas Retina Associates, Arlington, Texas
  - Retina Research Center, Austin, Texas
  - Strategic Clinical Research Group, LLC, Willow Park, Texas
  - Retina Associates of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Khanani AM, Patel SS, Ferrone PJ, Osborne A, Sahni J, Grzeschik S, Basu K, Ehrlich JS, Haskova Z, Dugel PU. Efficacy of Every Four Monthly and Quarterly Dosing of Faricimab vs Ranibizumab in Neovascular Age-Related Macular Degeneration: The STAIRWAY Phase 2 Randomized Clinical Trial. JAMA Ophthalmol. 2020 Sep 1;138(9):964-972. doi: 10.1001/jamaophthalmol.2020.2699. PMID 32729897

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 6 mg Faricimab Q12W | 6 mg Faricimab Q16W | 0.5 mg Ranibizumab Q4W
Started | 24 | 31 | 16
Completed | 21 | 28 | 16
Not Completed | 3 | 3 | 0
Not completed — Death | 1 | 2 | 0
Not completed — Physician Decision | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The efficacy population includes randomized participants grouped according to their assigned treatment. A total of 76 patients were randomized in the study, but 5 participants in total (all randomized to the 6 mg Faricimab Q12W Arm) were excluded from the analysis populations because of Good Clinical Practice (GCP) violations at a single site.
Groups:
- Total: Total of all reporting groups
Arm/Group | 6 mg Faricimab Q12W | 6 mg Faricimab Q16W | 0.5 mg Ranibizumab Q4W | Total
Number analyzed (Participants) | 24 | 31 | 16 | 71
Age, Continuous [Mean (Standard Deviation); unit: Years] | 80.3 (7.23) | 77.7 (8.38) | 77.3 (10.29) | 78.5 (8.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 18 | 10 | 41
  Male | 11 | 13 | 6 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 23 | 31 | 16 | 70
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 0 | 1
  Black or African American | 1 | 0 | 0 | 1
  White | 23 | 30 | 16 | 69
Best Corrected Visual Acuity (BCVA) Letter Score in the Study Eye at Baseline [Mean (Standard Deviation); unit: ETDRS Letters] — Best corrected visual acuity (BCVA) at a starting test distance of 4 meters was measured using a set of three Precision VisionTM or Lighthouse distance acuity charts (modified ETDRS Charts 1, 2, and R). The BCVA letter score ranges from 0 to 100 (best score attainable), with a higher score indicating better visual acuity.
  ETDRS Letters | 57.8 (10.46) | 60.4 (10.80) | 55.3 (12.08) | 58.4 (11.02)
Choroidal Neovascularization (CNV) Lesion Type in the Study Eye at Baseline [Count of Participants; unit: Participants]
  Classic and Occult CNV | 0 | 2 | 2 | 4
  Classic CNV | 9 | 9 | 6 | 24
  Occult CNV | 15 | 20 | 8 | 43
Central Foveal Thickness in the Study Eye at Baseline [Mean (Standard Deviation); unit: microns (μm)] — Central foveal thickness (CFT) was defined as the thickness from the inner limiting membrane to the retinal pigment epithelial at the horizontal slice closest to the center of the fovea, and it was measured using spectral domain optical coherence tomography (SD-OCT).
  microns (μm) | 290.8 (118.61) | 280.8 (98.95) | 375.6 (159.41) | 305.6 (125.42)
Central Subfield Thickness in the Study Eye at Baseline [Mean (Standard Deviation); unit: microns (μm)] — Central subfield thickness (CST) was defined as the mean thickness from the inner limiting membrane to the retinal pigment epithelial over the 1 millimetre (mm) central subfield, and it was measured using spectral domain optical coherence tomography (SD-OCT).
  microns (μm) | 417.9 (84.28) | 382.2 (80.87) | 443.1 (125.00) | 408.0 (95.36)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Best Corrected Visual Acuity (BCVA) at Week 40, Using the Early Treatment Diabetic Retinopathy Study (ETDRS) BCVA Charts
Description: Best corrected visual acuity (BCVA) at a starting test distance of 4 meters was measured using a set of three Precision VisionTM or Lighthouse distance acuity charts (modified ETDRS Charts 1, 2, and R) prior to dilating eyes by a trained and certified visual acuity examiner. The BCVA examiner was masked to study eye and treatment assignment and only performed the refraction and BCVA assessment. The BCVA examiner was also masked to the BCVA letter scores of a participant's previous visits and could only know the refraction data from previous visits. The BCVA letter score ranges from 0 to 100 (best score attainable), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity. The analysis was performed using a Mixed Model for Repeated Measurement (MMRM) model, which included an unstructured covariance and the categorical covariates of treatment group, visit, and visit by treatment group interaction and the continuous covariate of baseline BCVA.
Time Frame: Baseline, Week 40
Population: Efficacy population: participants grouped according to their assigned treatment.
Measure: Least Squares Mean (80% Confidence Interval); unit: ETDRS Letters
Arm/Group | 6 mg Faricimab Q12W | 6 mg Faricimab Q16W | 0.5 mg Ranibizumab Q4W
Number analyzed (Participants) | 24 | 31 | 16
ETDRS Letters | 9.3 [6.4 to 12.3] | 12.5 [9.9 to 15.1] | 11.4 [7.8 to 15.0]
Statistical Analysis 1: Comparison: 6 mg Faricimab Q12W vs 0.5 mg Ranibizumab Q4W; Test type: Other — The focus of this trial was estimation rather than hypothesis testing; Mean Difference (Net) = -2.1, 80% CI 2-sided [-6.8 to 2.6] — The difference was calculated as Faricimab Q12W arm minus Ranibizumab Q4W arm
Statistical Analysis 2: Comparison: 6 mg Faricimab Q16W vs 0.5 mg Ranibizumab Q4W; Test type: Other — The focus of this trial was estimation rather than hypothesis testing; Mean Difference (Net) = 1.1, 80% CI 2-sided [-3.4 to 5.5] — The difference was calculated as Faricimab Q16W arm minus Ranibizumab Q4W arm

2. Secondary Outcome: Mean Change From Baseline in BCVA at Specified Timepoints, Using the ETDRS BCVA Charts
Description: as for outcome 1
Time Frame: Baseline, Day 7, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: Efficacy population: participants grouped according to their assigned treatment.
Measure: Least Squares Mean (80% Confidence Interval); unit: ETDRS Letters
Arm/Group | 6 mg Faricimab Q12W | 6 mg Faricimab Q16W | 0.5 mg Ranibizumab Q4W
Number analyzed (Participants) | 24 | 31 | 16
ETDRS Letters
  Day 7 | 3.78 [2.33 to 5.24] | 4.62 [3.33 to 5.91] | 3.53 [1.74 to 5.33]
  Week 4 | 5.99 [4.10 to 7.88] | 7.55 [5.88 to 9.22] | 7.53 [5.21 to 9.86]
  Week 8 | 5.28 [2.88 to 7.69] | 9.15 [7.01 to 11.29] | 10.55 [7.55 to 13.54]
  Week 12 | 7.31 [4.87 to 9.75] | 10.19 [8.04 to 12.34] | 9.91 [6.94 to 12.88]
  Week 16 | 8.31 [5.93 to 10.68] | 11.62 [9.52 to 13.71] | 10.78 [7.89 to 13.68]
  Week 20 | 8.02 [5.35 to 10.69] | 10.40 [8.05 to 12.76] | 11.53 [8.28 to 14.78]
  Week 24 | 8.11 [5.53 to 10.69] | 10.37 [8.10 to 12.65] | 10.97 [7.83 to 14.11]
  Week 28 | 9.59 [7.06 to 12.12] | 11.82 [9.59 to 14.05] | 12.16 [9.08 to 15.23]
  Week 32 | 9.87 [7.21 to 12.53] | 12.44 [10.10 to 14.79] | 11.91 [8.67 to 15.14]
  Week 36 | 9.01 [6.14 to 11.87] | 12.38 [9.86 to 14.90] | 12.03 [8.57 to 15.50]
  Week 40 | 9.33 [6.37 to 12.29] | 12.47 [9.86 to 15.08] | 11.42 [7.83 to 15.01]
  Week 44 | 9.38 [6.42 to 12.34] | 12.07 [9.48 to 14.67] | 11.22 [7.65 to 14.79]
  Week 48 | 9.53 [6.51 to 12.55] | 10.99 [8.33 to 13.64] | 10.22 [6.57 to 13.86]
  Week 52 | 10.08 [7.05 to 13.12] | 11.42 [8.75 to 14.09] | 9.59 [5.93 to 13.25]
Statistical Analysis 1: Comparison: 6 mg Faricimab Q12W vs 0.5 mg Ranibizumab Q4W; Week 40: Faricimab Q12W vs. Ranibizumab Q4W; Test type: Other — The focus of this trial was estimation rather than hypothesis testing; Mean Difference (Net) = -2.09, 80% CI 2-sided [-6.75 to 2.56] — The difference was calculated as Faricimab Q12W arm minus Ranibizumab Q4W arm
Statistical Analysis 2: Comparison: 6 mg Faricimab Q16W vs 0.5 mg Ranibizumab Q4W; Week 40: Faricimab Q16W vs. Ranibizumab Q4W; Test type: Other — The focus of this trial was estimation rather than hypothesis testing; Mean Difference (Net) = 1.05, 80% CI 2-sided [-3.40 to 5.49] — The difference was calculated as Faricimab Q16W arm minus Ranibizumab Q4W arm
Statistical Analysis 3: Comparison: 6 mg Faricimab Q12W vs 0.5 mg Ranibizumab Q4W; Week 52: Faricimab Q12W vs. Ranibizumab Q4W; Test type: Other — The focus of this trial was estimation rather than hypothesis testing; Mean Difference (Net) = 0.49, 80% CI 2-sided [-4.26 to 5.25] — The difference was calculated as Faricimab Q12W arm minus Ranibizumab Q4W arm
Statistical Analysis 4: Comparison: 6 mg Faricimab Q16W vs 0.5 mg Ranibizumab Q4W; Week 52: Faricimab Q16W vs. Ranibizumab Q4W; Test type: Other — The focus of this trial was estimation rather than hypothesis testing; Mean Difference (Net) = 1.83, 80% CI 2-sided [-2.71 to 6.37] — The difference was calculated as Faricimab Q16W arm minus Ranibizumab Q4W arm

3. Secondary Outcome: Number and Percentage of Participants Gaining Greater Than or Equal to (≥)15, ≥10, ≥5, or ≥0 Letters From Baseline in BCVA at Specified Timepoints
Description: Best corrected visual acuity (BCVA) at a starting test distance of 4 meters was measured using a set of three Precision VisionTM or Lighthouse distance acuity charts (modified ETDRS Charts 1, 2, and R) prior to dilating eyes by a trained and certified visual acuity examiner. The BCVA examiner was masked to study eye and treatment assignment and only performed the refraction and BCVA assessment. The BCVA examiner was also masked to the BCVA letter scores of a participant's previous visits and could only know the refraction data from previous visits. The BCVA letter score ranges from 0 to 100 (best score attainable), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity. This analysis was performed on observed data.
Time Frame: Baseline, Day 7, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: Efficacy population: participants grouped according to their assigned treatment. This analysis of observed data included participants with non-missing assessments at each timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | 6 mg Faricimab Q12W | 6 mg Faricimab Q16W | 0.5 mg Ranibizumab Q4W
Number analyzed (Participants) | 24 | 31 | 16
Participants
  Day 7: Gaining ≥15 Letters | 1 | 2 | 1
  Day 7: Gaining ≥10 Letters | 2 | 4 | 1
  Day 7: Gaining ≥5 Letters | 11 | 16 | 6
  Day 7: Gaining ≥0 Letters | 20 | 26 | 15
  Week 4: Gaining ≥15 Letters | 3 | 4 | 3
  Week 4: Gaining ≥10 Letters | 5 | 8 | 5
  Week 4: Gaining ≥5 Letters | 15 | 19 | 8
  Week 4: Gaining ≥0 Letters | 20 | 30 | 15
  Week 8: Gaining ≥15 Letters: number analyzed (Participants) | 24 | 30 | 15
  Week 8: Gaining ≥15 Letters | 3 | 5 | 6
  Week 8: Gaining ≥10 Letters: number analyzed (Participants) | 24 | 30 | 15
  Week 8: Gaining ≥10 Letters | 7 | 10 | 8
  Week 8: Gaining ≥5 Letters: number analyzed (Participants) | 24 | 30 | 15
  Week 8: Gaining ≥5 Letters | 14 | 26 | 10
  Week 8: Gaining ≥0 Letters: number analyzed (Participants) | 24 | 30 | 15
  Week 8: Gaining ≥0 Letters | 21 | 28 | 15
  Week 12: Gaining ≥15 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 12: Gaining ≥15 Letters | 2 | 7 | 3
  Week 12: Gaining ≥10 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 12: Gaining ≥10 Letters | 8 | 16 | 7
  Week 12: Gaining ≥5 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 12: Gaining ≥5 Letters | 15 | 23 | 11
  Week 12: Gaining ≥0 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 12: Gaining ≥0 Letters | 19 | 29 | 15
  Week 16: Gaining ≥15 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 16: Gaining ≥15 Letters | 4 | 9 | 3
  Week 16: Gaining ≥10 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 16: Gaining ≥10 Letters | 10 | 16 | 8
  Week 16: Gaining ≥5 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 16: Gaining ≥5 Letters | 16 | 27 | 13
  Week 16: Gaining ≥0 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 16: Gaining ≥0 Letters | 21 | 29 | 16
  Week 20: Gaining ≥15 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 20: Gaining ≥15 Letters | 4 | 10 | 3
  Week 20: Gaining ≥10 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 20: Gaining ≥10 Letters | 10 | 17 | 9
  Week 20: Gaining ≥5 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 20: Gaining ≥5 Letters | 16 | 22 | 14
  Week 20: Gaining ≥0 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 20: Gaining ≥0 Letters | 20 | 26 | 16
  Week 24: Gaining ≥15 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 24: Gaining ≥15 Letters | 4 | 8 | 4
  Week 24: Gaining ≥10 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 24: Gaining ≥10 Letters | 9 | 16 | 9
  Week 24: Gaining ≥5 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 24: Gaining ≥5 Letters | 15 | 22 | 12
  Week 24: Gaining ≥0 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 24: Gaining ≥0 Letters | 19 | 27 | 15
  Week 28: Gaining ≥15 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 28: Gaining ≥15 Letters | 6 | 12 | 5
  Week 28: Gaining ≥10 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 28: Gaining ≥10 Letters | 13 | 15 | 9
  Week 28: Gaining ≥5 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 28: Gaining ≥5 Letters | 16 | 24 | 11
  Week 28: Gaining ≥0 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 28: Gaining ≥0 Letters | 21 | 27 | 16
  Week 32: Gaining ≥15 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 32: Gaining ≥15 Letters | 7 | 11 | 6
  Week 32: Gaining ≥10 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 32: Gaining ≥10 Letters | 11 | 18 | 9
  Week 32: Gaining ≥5 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 32: Gaining ≥5 Letters | 17 | 27 | 11
  Week 32: Gaining ≥0 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 32: Gaining ≥0 Letters | 22 | 28 | 15
  Week 36: Gaining ≥15 Letters: number analyzed (Participants) | 22 | 29 | 16
  Week 36: Gaining ≥15 Letters | 7 | 11 | 6
  Week 36: Gaining ≥10 Letters: number analyzed (Participants) | 22 | 29 | 16
  Week 36: Gaining ≥10 Letters | 10 | 20 | 10
  Week 36: Gaining ≥5 Letters: number analyzed (Participants) | 22 | 29 | 16
  Week 36: Gaining ≥5 Letters | 15 | 24 | 12
  Week 36: Gaining ≥0 Letters: number analyzed (Participants) | 22 | 29 | 16
  Week 36: Gaining ≥0 Letters | 19 | 25 | 15
  Week 40: Gaining ≥15 Letters: number analyzed (Participants) | 21 | 28 | 15
  Week 40: Gaining ≥15 Letters | 8 | 11 | 5
  Week 40: Gaining ≥10 Letters: number analyzed (Participants) | 21 | 28 | 15
  Week 40: Gaining ≥10 Letters | 11 | 18 | 8
  Week 40: Gaining ≥5 Letters: number analyzed (Participants) | 21 | 28 | 15
  Week 40: Gaining ≥5 Letters | 15 | 24 | 10
  Week 40: Gaining ≥0 Letters: number analyzed (Participants) | 21 | 28 | 15
  Week 40: Gaining ≥0 Letters | 17 | 27 | 13
  Week 44: Gaining ≥15 Letters: number analyzed (Participants) | 20 | 29 | 16
  Week 44: Gaining ≥15 Letters | 7 | 13 | 6
  Week 44: Gaining ≥10 Letters: number analyzed (Participants) | 20 | 29 | 16
  Week 44: Gaining ≥10 Letters | 12 | 15 | 9
  Week 44: Gaining ≥5 Letters: number analyzed (Participants) | 20 | 29 | 16
  Week 44: Gaining ≥5 Letters | 13 | 26 | 11
  Week 44: Gaining ≥0 Letters: number analyzed (Participants) | 20 | 29 | 16
  Week 44: Gaining ≥0 Letters | 15 | 27 | 13
  Week 48: Gaining ≥15 Letters: number analyzed (Participants) | 21 | 28 | 16
  Week 48: Gaining ≥15 Letters | 7 | 10 | 6
  Week 48: Gaining ≥10 Letters: number analyzed (Participants) | 21 | 28 | 16
  Week 48: Gaining ≥10 Letters | 12 | 17 | 10
  Week 48: Gaining ≥5 Letters: number analyzed (Participants) | 21 | 28 | 16
  Week 48: Gaining ≥5 Letters | 15 | 20 | 11
  Week 48: Gaining ≥0 Letters: number analyzed (Participants) | 21 | 28 | 16
  Week 48: Gaining ≥0 Letters | 18 | 26 | 12
  Week 52: Gaining ≥15 Letters: number analyzed (Participants) | 21 | 28 | 16
  Week 52: Gaining ≥15 Letters | 7 | 13 | 6
  Week 52: Gaining ≥10 Letters: number analyzed (Participants) | 21 | 28 | 16
  Week 52: Gaining ≥10 Letters | 11 | 17 | 9
  Week 52: Gaining ≥5 Letters: number analyzed (Participants) | 21 | 28 | 16
  Week 52: Gaining ≥5 Letters | 14 | 23 | 9
  Week 52: Gaining ≥0 Letters: number analyzed (Participants) | 21 | 28 | 16
  Week 52: Gaining ≥0 Letters | 17 | 26 | 13

4. Secondary Outcome: Percentage of Participants Gaining ≥15 Letters From Baseline in BCVA at Specified Timepoints
Description: Best corrected visual acuity (BCVA) at a starting test distance of 4 meters was measured using a set of three Precision VisionTM or Lighthouse distance acuity charts (modified ETDRS Charts 1, 2, and R) prior to dilating eyes by a trained and certified visual acuity examiner. The BCVA examiner was masked to study eye and treatment assignment and only performed the refraction and BCVA assessment. The BCVA examiner was also masked to the BCVA letter scores of a participant's previous visits and could only know the refraction data from previous visits. The BCVA letter score ranges from 0 to 100 (best score attainable), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity. This analysis was performed on observed data. The 80% confidence intervals were calculated using the Wald method.
Time Frame: Baseline, Day 7, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: as for outcome 3
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | 6 mg Faricimab Q12W | 6 mg Faricimab Q16W | 0.5 mg Ranibizumab Q4W
Number analyzed (Participants) | 24 | 31 | 16
Percentage of participants
  Day 7 | 4.2 [0.00 to 9.39] | 6.5 [0.80 to 12.11] | 6.3 [0.00 to 14.01]
  Week 4 | 12.5 [3.85 to 21.15] | 12.9 [5.19 to 20.62] | 18.8 [6.24 to 31.26]
  Week 8: number analyzed (Participants) | 24 | 30 | 15
  Week 8 | 12.5 [3.85 to 21.15] | 16.7 [7.95 to 25.39] | 40.0 [23.79 to 56.21]
  Week 12: number analyzed (Participants) | 23 | 30 | 16
  Week 12 | 8.7 [1.17 to 16.23] | 23.3 [13.44 to 33.23] | 18.8 [6.24 to 31.26]
  Week 16: number analyzed (Participants) | 23 | 30 | 16
  Week 16 | 17.4 [7.26 to 27.52] | 30.0 [19.28 to 40.72] | 18.8 [6.24 to 31.26]
  Week 20: number analyzed (Participants) | 23 | 30 | 16
  Week 20 | 17.4 [7.26 to 27.52] | 33.3 [22.30 to 44.36] | 18.8 [6.24 to 31.26]
  Week 24: number analyzed (Participants) | 23 | 30 | 16
  Week 24 | 17.4 [7.26 to 27.52] | 26.7 [16.32 to 37.01] | 25.0 [11.13 to 38.87]
  Week 28: number analyzed (Participants) | 23 | 30 | 16
  Week 28 | 26.1 [14.35 to 37.82] | 40.0 [28.54 to 51.46] | 31.3 [16.40 to 46.10]
  Week 32: number analyzed (Participants) | 23 | 30 | 16
  Week 32 | 30.4 [18.14 to 42.73] | 36.7 [25.39 to 47.94] | 37.5 [21.99 to 53.01]
  Week 36: number analyzed (Participants) | 22 | 29 | 16
  Week 36 | 31.8 [19.09 to 44.54] | 37.9 [26.38 to 49.48] | 37.5 [21.99 to 53.01]
  Week 40: number analyzed (Participants) | 21 | 28 | 15
  Week 40 | 38.1 [24.51 to 51.68] | 39.3 [27.46 to 51.11] | 33.3 [17.73 to 48.93]
  Week 44: number analyzed (Participants) | 20 | 29 | 16
  Week 44 | 35.0 [21.33 to 48.67] | 44.8 [32.99 to 56.66] | 37.5 [21.99 to 53.01]
  Week 48: number analyzed (Participants) | 21 | 28 | 16
  Week 48 | 33.3 [20.15 to 46.52] | 35.7 [24.11 to 47.32] | 37.5 [21.99 to 53.01]
  Week 52: number analyzed (Participants) | 21 | 28 | 16
  Week 52 | 33.3 [20.15 to 46.52] | 46.4 [34.35 to 58.51] | 37.5 [21.99 to 53.01]
Statistical Analysis 1: Comparison: 6 mg Faricimab Q12W vs 0.5 mg Ranibizumab Q4W; Week 40: Faricimab Q12W vs. Ranibizumab Q4W; Test type: Other — The focus of this trial was estimation rather than hypothesis testing; Difference in Percentage of Participants = 4.76, 80% CI 2-sided [-15.92 to 25.44] — The difference was calculated as Faricimab Q12W arm minus Ranibizumab Q4W arm
Statistical Analysis 2: Comparison: 6 mg Faricimab Q16W vs 0.5 mg Ranibizumab Q4W; Week 40: Faricimab Q16W vs. Ranibizumab Q4W; Test type: Other — The focus of this trial was estimation rather than hypothesis testing; Difference in Percentage of Participants = 5.95, 80% CI 2-sided [-13.62 to 25.53] — The difference was calculated as Faricimab Q16W arm minus Ranibizumab Q4W arm
Statistical Analysis 3: Comparison: 6 mg Faricimab Q12W vs 0.5 mg Ranibizumab Q4W; Week 52: Faricimab Q12W vs. Ranibizumab Q4W; Test type: Other — The focus of this trial was estimation rather than hypothesis testing; Difference in Percentage of Participants = -4.17, 80% CI 2-sided [-24.52 to 16.19] — The difference was calculated as Faricimab Q12W arm minus Ranibizumab Q4W arm
Statistical Analysis 4: Comparison: 6 mg Faricimab Q16W vs 0.5 mg Ranibizumab Q4W; Week 52: Faricimab Q16W vs. Ranibizumab Q4W; Test type: Other — The focus of this trial was estimation rather than hypothesis testing; Difference in Percentage of Participants = 8.93, 80% CI 2-sided [-10.73 to 28.59] — The difference was calculated as Faricimab Q16W arm minus Ranibizumab Q4W arm

5. Secondary Outcome: Number and Percentage of Participants Not Losing ≥15, ≥10, ≥5, or ≥0 Letters From Baseline in BCVA at Specified Timepoints
Description: Best corrected visual acuity (BCVA) at a starting test distance of 4 meters was measured using a set of three Precision VisionTM or Lighthouse distance acuity charts (modified ETDRS Charts 1, 2, and R) prior to dilating eyes by a trained and certified visual acuity examiner. The BCVA examiner was masked to study eye and treatment assignment and only performed the refraction and BCVA assessment. The BCVA examiner was also masked to the BCVA letter scores of a participant's previous visits and could only know the refraction data from previous visits. The BCVA letter score ranges from 0 to 100 (best score attainable), and a loss in BCVA letter score from baseline indicates worsening in visual acuity. This analysis was performed on observed data.
Time Frame: Baseline, Day 7, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | 6 mg Faricimab Q12W | 6 mg Faricimab Q16W | 0.5 mg Ranibizumab Q4W
Number analyzed (Participants) | 24 | 31 | 16
Participants
  Day 7: Not Losing ≥15 Letters | 24 | 31 | 16
  Day 7: Not Losing ≥10 Letters | 24 | 31 | 16
  Day 7: Not Losing ≥5 Letters | 21 | 29 | 15
  Day 7: Not Losing ≥0 Letters | 18 | 24 | 10
  Week 4: Not Losing ≥15 Letters | 24 | 31 | 16
  Week 4: Not Losing ≥10 Letters | 24 | 31 | 16
  Week 4: Not Losing ≥5 Letters | 23 | 31 | 16
  Week 4: Not Losing ≥0 Letters | 18 | 29 | 13
  Week 8: Not Losing ≥15 Letters: number analyzed (Participants) | 24 | 30 | 15
  Week 8: Not Losing ≥15 Letters | 23 | 30 | 15
  Week 8: Not Losing ≥10 Letters: number analyzed (Participants) | 24 | 30 | 15
  Week 8: Not Losing ≥10 Letters | 23 | 30 | 15
  Week 8: Not Losing ≥5 Letters: number analyzed (Participants) | 24 | 30 | 15
  Week 8: Not Losing ≥5 Letters | 22 | 29 | 15
  Week 8: Not Losing ≥0 Letters: number analyzed (Participants) | 24 | 30 | 15
  Week 8: Not Losing ≥0 Letters | 20 | 28 | 13
  Week 12: Not Losing ≥15 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 12: Not Losing ≥15 Letters | 23 | 29 | 16
  Week 12: Not Losing ≥10 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 12: Not Losing ≥10 Letters | 23 | 29 | 16
  Week 12: Not Losing ≥5 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 12: Not Losing ≥5 Letters | 23 | 29 | 16
  Week 12: Not Losing ≥0 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 12: Not Losing ≥0 Letters | 19 | 28 | 14
  Week 16: Not Losing ≥15 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 16: Not Losing ≥15 Letters | 23 | 29 | 16
  Week 16: Not Losing ≥10 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 16: Not Losing ≥10 Letters | 23 | 29 | 16
  Week 16: Not Losing ≥5 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 16: Not Losing ≥5 Letters | 22 | 29 | 16
  Week 16: Not Losing ≥0 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 16: Not Losing ≥0 Letters | 19 | 29 | 16
  Week 20: Not Losing ≥15 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 20: Not Losing ≥15 Letters | 23 | 29 | 16
  Week 20: Not Losing ≥10 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 20: Not Losing ≥10 Letters | 23 | 29 | 16
  Week 20: Not Losing ≥5 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 20: Not Losing ≥5 Letters | 22 | 29 | 16
  Week 20: Not Losing ≥0 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 20: Not Losing ≥0 Letters | 19 | 24 | 14
  Week 24: Not Losing ≥15 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 24: Not Losing ≥15 Letters | 23 | 30 | 16
  Week 24: Not Losing ≥10 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 24: Not Losing ≥10 Letters | 22 | 29 | 16
  Week 24: Not Losing ≥5 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 24: Not Losing ≥5 Letters | 22 | 28 | 16
  Week 24: Not Losing ≥0 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 24: Not Losing ≥0 Letters | 19 | 27 | 14
  Week 28: Not Losing ≥15 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 28: Not Losing ≥15 Letters | 23 | 29 | 16
  Week 28: Not Losing ≥10 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 28: Not Losing ≥10 Letters | 23 | 28 | 16
  Week 28: Not Losing ≥5 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 28: Not Losing ≥5 Letters | 21 | 28 | 16
  Week 28: Not Losing ≥0 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 28: Not Losing ≥0 Letters | 20 | 27 | 16
  Week 32: Not Losing ≥15 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 32: Not Losing ≥15 Letters | 23 | 29 | 16
  Week 32: Not Losing ≥10 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 32: Not Losing ≥10 Letters | 23 | 28 | 16
  Week 32: Not Losing ≥5 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 32: Not Losing ≥5 Letters | 22 | 28 | 16
  Week 32: Not Losing ≥0 Letters: number analyzed (Participants) | 23 | 30 | 16
  Week 32: Not Losing ≥0 Letters | 20 | 28 | 13
  Week 36: Not Losing ≥15 Letters: number analyzed (Participants) | 22 | 29 | 16
  Week 36: Not Losing ≥15 Letters | 21 | 28 | 16
  Week 36: Not Losing ≥10 Letters: number analyzed (Participants) | 22 | 29 | 16
  Week 36: Not Losing ≥10 Letters | 21 | 28 | 16
  Week 36: Not Losing ≥5 Letters: number analyzed (Participants) | 22 | 29 | 16
  Week 36: Not Losing ≥5 Letters | 20 | 27 | 15
  Week 36: Not Losing ≥0 Letters: number analyzed (Participants) | 22 | 29 | 16
  Week 36: Not Losing ≥0 Letters | 19 | 25 | 14
  Week 40: Not Losing ≥15 Letters: number analyzed (Participants) | 21 | 28 | 15
  Week 40: Not Losing ≥15 Letters | 20 | 27 | 15
  Week 40: Not Losing ≥10 Letters: number analyzed (Participants) | 21 | 28 | 15
  Week 40: Not Losing ≥10 Letters | 20 | 27 | 15
  Week 40: Not Losing ≥5 Letters: number analyzed (Participants) | 21 | 28 | 15
  Week 40: Not Losing ≥5 Letters | 19 | 27 | 15
  Week 40: Not Losing ≥0 Letters: number analyzed (Participants) | 21 | 28 | 15
  Week 40: Not Losing ≥0 Letters | 17 | 25 | 12
  Week 44: Not Losing ≥15 Letters: number analyzed (Participants) | 20 | 29 | 16
  Week 44: Not Losing ≥15 Letters | 20 | 28 | 16
  Week 44: Not Losing ≥10 Letters: number analyzed (Participants) | 20 | 29 | 16
  Week 44: Not Losing ≥10 Letters | 20 | 28 | 16
  Week 44: Not Losing ≥5 Letters: number analyzed (Participants) | 20 | 29 | 16
  Week 44: Not Losing ≥5 Letters | 17 | 28 | 16
  Week 44: Not Losing ≥0 Letters: number analyzed (Participants) | 20 | 29 | 16
  Week 44: Not Losing ≥0 Letters | 14 | 27 | 12
  Week 48: Not Losing ≥15 Letters: number analyzed (Participants) | 21 | 28 | 16
  Week 48: Not Losing ≥15 Letters | 21 | 27 | 16
  Week 48: Not Losing ≥10 Letters: number analyzed (Participants) | 21 | 28 | 16
  Week 48: Not Losing ≥10 Letters | 20 | 27 | 16
  Week 48: Not Losing ≥5 Letters: number analyzed (Participants) | 21 | 28 | 16
  Week 48: Not Losing ≥5 Letters | 19 | 27 | 15
  Week 48: Not Losing ≥0 Letters: number analyzed (Participants) | 21 | 28 | 16
  Week 48: Not Losing ≥0 Letters | 16 | 25 | 11
  Week 52: Not Losing ≥15 Letters: number analyzed (Participants) | 21 | 28 | 16
  Week 52: Not Losing ≥15 Letters | 21 | 27 | 16
  Week 52: Not Losing ≥10 Letters: number analyzed (Participants) | 21 | 28 | 16
  Week 52: Not Losing ≥10 Letters | 21 | 27 | 16
  Week 52: Not Losing ≥5 Letters: number analyzed (Participants) | 21 | 28 | 16
  Week 52: Not Losing ≥5 Letters | 20 | 27 | 15
  Week 52: Not Losing ≥0 Letters: number analyzed (Participants) | 21 | 28 | 16
  Week 52: Not Losing ≥0 Letters | 16 | 26 | 11

6. Secondary Outcome: Percentage of Participants Not Losing ≥15 Letters From Baseline in BCVA at Specified Timepoints
Description: as for outcome 4
Time Frame: Baseline, Day 7, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: as for outcome 3
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | 6 mg Faricimab Q12W | 6 mg Faricimab Q16W | 0.5 mg Ranibizumab Q4W
Number analyzed (Participants) | 24 | 31 | 16
Percentage of participants
  Day 7 | 100.0 [100.00 to 100.00] | 100.0 [100.00 to 100.00] | 100.0 [100.00 to 100.00]
  Week 4 | 100.0 [100.00 to 100.00] | 100.0 [100.00 to 100.00] | 100.0 [100.00 to 100.00]
  Week 8: number analyzed (Participants) | 24 | 30 | 15
  Week 8 | 95.8 [90.61 to 100.00] | 100.0 [100.00 to 100.00] | 100.0 [100.00 to 100.00]
  Week 12: number analyzed (Participants) | 23 | 30 | 16
  Week 12 | 100.0 [100.00 to 100.00] | 96.7 [92.47 to 100.00] | 100.0 [100.00 to 100.00]
  Week 16: number analyzed (Participants) | 23 | 30 | 16
  Week 16 | 100.0 [100.00 to 100.00] | 96.7 [92.47 to 100.00] | 100.0 [100.00 to 100.00]
  Week 20: number analyzed (Participants) | 23 | 30 | 16
  Week 20 | 100.0 [100.00 to 100.00] | 96.7 [92.47 to 100.00] | 100.0 [100.00 to 100.00]
  Week 24: number analyzed (Participants) | 23 | 30 | 16
  Week 24 | 100.0 [100.00 to 100.00] | 100.0 [100.00 to 100.00] | 100.0 [100.00 to 100.00]
  Week 28: number analyzed (Participants) | 23 | 30 | 16
  Week 28 | 100.0 [100.00 to 100.00] | 96.7 [92.47 to 100.00] | 100.0 [100.00 to 100.00]
  Week 32: number analyzed (Participants) | 23 | 30 | 16
  Week 32 | 100.0 [100.00 to 100.00] | 96.7 [92.47 to 100.00] | 100.0 [100.00 to 100.00]
  Week 36: number analyzed (Participants) | 22 | 29 | 16
  Week 36 | 95.5 [89.76 to 100.00] | 96.6 [92.21 to 100.00] | 100.0 [100.00 to 100.00]
  Week 40: number analyzed (Participants) | 21 | 28 | 15
  Week 40 | 95.2 [89.28 to 100.00] | 96.4 [91.93 to 100.00] | 100.0 [100.00 to 100.00]
  Week 44: number analyzed (Participants) | 20 | 29 | 16
  Week 44 | 100.0 [100.00 to 100.00] | 96.6 [92.21 to 100.00] | 100.0 [100.00 to 100.00]
  Week 48: number analyzed (Participants) | 21 | 28 | 16
  Week 48 | 100.0 [100.00 to 100.00] | 96.4 [91.93 to 100.00] | 100.0 [100.00 to 100.00]
  Week 52: number analyzed (Participants) | 21 | 28 | 16
  Week 52 | 100.0 [100.00 to 100.00] | 96.4 [91.93 to 100.00] | 100.0 [100.00 to 100.00]
Statistical Analysis 1: Comparison: 6 mg Faricimab Q12W vs 0.5 mg Ranibizumab Q4W; Week 40: Faricimab Q12W vs. Ranibizumab Q4W; Test type: Other — The focus of this trial was estimation rather than hypothesis testing; Difference in Percentage of Participants = -4.76, 80% CI 2-sided [-10.72 to 1.19] — The difference was calculated as Faricimab Q12W arm minus Ranibizumab Q4W arm
Statistical Analysis 2: Comparison: 6 mg Faricimab Q16W vs 0.5 mg Ranibizumab Q4W; Week 40: Faricimab Q16W vs. Ranibizumab Q4W; Test type: Other — The focus of this trial was estimation rather than hypothesis testing; Difference in Percentage of Participants = -3.57, 80% CI 2-sided [-8.07 to 0.92] — The difference was calculated as Faricimab Q16W arm minus Ranibizumab Q4W arm
Statistical Analysis 3: Comparison: 6 mg Faricimab Q12W vs 0.5 mg Ranibizumab Q4W; Week 52: Faricimab Q12W vs. Ranibizumab Q4W; Test type: Other — The focus of this trial was estimation rather than hypothesis testing; Difference in Percentage of Participants = 0 — The difference was calculated as Faricimab Q12W arm minus Ranibizumab Q4W arm
Statistical Analysis 4: Comparison: 6 mg Faricimab Q16W vs 0.5 mg Ranibizumab Q4W; Week 52: Faricimab Q16W vs. Ranibizumab Q4W; Test type: Other — The focus of this trial was estimation rather than hypothesis testing; Difference in Percentage of Participants = -3.57, 80% CI 2-sided [-8.07 to 0.92] — The difference was calculated as Faricimab Q16W arm minus Ranibizumab Q4W arm

7. Secondary Outcome: Percentage of Participants With BCVA Snellen Equivalent of 20/40 or Better at Specified Timepoints
Description: as for outcome 4
Time Frame: Baseline, Day 7, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: as for outcome 3
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | 6 mg Faricimab Q12W | 6 mg Faricimab Q16W | 0.5 mg Ranibizumab Q4W
Number analyzed (Participants) | 24 | 31 | 16
Percentage of participants
  Baseline | 12.5 [3.85 to 21.15] | 22.6 [12.96 to 32.20] | 18.8 [6.24 to 31.26]
  Day 7 | 20.8 [10.21 to 31.46] | 45.2 [33.71 to 56.62] | 18.8 [6.24 to 31.26]
  Week 4 | 45.8 [32.80 to 58.87] | 51.6 [40.11 to 63.12] | 25.0 [11.13 to 38.87]
  Week 8: number analyzed (Participants) | 24 | 30 | 15
  Week 8 | 41.7 [28.77 to 54.56] | 70.0 [59.28 to 80.72] | 20.0 [6.76 to 33.24]
  Week 12: number analyzed (Participants) | 23 | 30 | 16
  Week 12 | 43.5 [30.23 to 56.73] | 73.3 [62.99 to 83.68] | 31.3 [16.40 to 46.10]
  Week 16: number analyzed (Participants) | 23 | 30 | 16
  Week 16 | 52.2 [38.83 to 65.52] | 70.0 [59.28 to 80.72] | 43.8 [27.86 to 59.64]
  Week 20: number analyzed (Participants) | 23 | 30 | 16
  Week 20 | 47.8 [34.48 to 61.17] | 73.3 [62.99 to 83.68] | 50.0 [33.98 to 66.02]
  Week 24: number analyzed (Participants) | 23 | 30 | 16
  Week 24 | 56.5 [43.27 to 69.77] | 70.0 [59.28 to 80.72] | 37.5 [21.99 to 53.01]
  Week 28: number analyzed (Participants) | 23 | 30 | 16
  Week 28 | 56.5 [43.27 to 69.77] | 73.3 [62.99 to 83.68] | 37.5 [21.99 to 53.01]
  Week 32: number analyzed (Participants) | 23 | 30 | 16
  Week 32 | 60.9 [47.83 to 73.91] | 70.0 [59.28 to 80.72] | 43.8 [27.86 to 59.64]
  Week 36: number analyzed (Participants) | 22 | 29 | 16
  Week 36 | 59.1 [45.66 to 72.52] | 75.9 [65.68 to 86.05] | 43.8 [27.86 to 59.64]
  Week 40: number analyzed (Participants) | 21 | 28 | 15
  Week 40 | 61.9 [48.32 to 75.49] | 78.6 [68.63 to 88.51] | 40.0 [23.79 to 56.21]
  Week 44: number analyzed (Participants) | 20 | 29 | 16
  Week 44 | 50.0 [35.67 to 64.33] | 72.4 [61.78 to 83.05] | 37.5 [21.99 to 53.01]
  Week 48: number analyzed (Participants) | 21 | 28 | 16
  Week 48 | 57.1 [43.30 to 70.98] | 75.0 [64.51 to 85.49] | 37.5 [21.99 to 53.01]
  Week 52: number analyzed (Participants) | 21 | 28 | 16
  Week 52 | 57.1 [43.30 to 70.98] | 71.4 [60.49 to 82.37] | 37.5 [21.99 to 53.01]
Statistical Analysis 1: Comparison: 6 mg Faricimab Q12W vs 0.5 mg Ranibizumab Q4W; Week 40: Faricimab Q12W vs. Ranibizumab Q4W; Test type: Other — The focus of this trial was estimation rather than hypothesis testing; Difference in Percentage of Participants = 21.90, 80% CI 2-sided [0.76 to 43.05] — The difference was calculated as Faricimab Q12W arm minus Ranibizumab Q4W arm
Statistical Analysis 2: Comparison: 6 mg Faricimab Q16W vs 0.5 mg Ranibizumab Q4W; Week 40: Faricimab Q16W vs. Ranibizumab Q4W; Test type: Other — The focus of this trial was estimation rather than hypothesis testing; Difference in Percentage of Participants = 38.57, 80% CI 2-sided [19.56 to 57.59] — The difference was calculated as Faricimab Q16W arm minus Ranibizumab Q4W arm
Statistical Analysis 3: Comparison: 6 mg Faricimab Q12W vs 0.5 mg Ranibizumab Q4W; Week 52: Faricimab Q12W vs. Ranibizumab Q4W; Test type: Other — The focus of this trial was estimation rather than hypothesis testing; Difference in Percentage of Participants = 19.64, 80% CI 2-sided [-1.14 to 40.43] — The difference was calculated as Faricimab Q12W arm minus Ranibizumab Q4W arm
Statistical Analysis 4: Comparison: 6 mg Faricimab Q16W vs 0.5 mg Ranibizumab Q4W; Week 52: Faricimab Q16W vs. Ranibizumab Q4W; Test type: Other — The focus of this trial was estimation rather than hypothesis testing; Difference in Percentage of Participants = 33.93, 80% CI 2-sided [14.95 to 52.91] — The difference was calculated as Faricimab Q16W arm minus Ranibizumab Q4W arm

8. Secondary Outcome: Percentage of Participants With BCVA Snellen Equivalent of 20/200 or Worse at Specified Timepoints
Description: as for outcome 4
Time Frame: Baseline, Day 7, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: as for outcome 3
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | 6 mg Faricimab Q12W | 6 mg Faricimab Q16W | 0.5 mg Ranibizumab Q4W
Number analyzed (Participants) | 24 | 31 | 16
Percentage of participants
  Baseline | 8.3 [1.10 to 15.56] | 3.2 [0.00 to 7.29] | 12.5 [1.90 to 23.10]
  Day 7 | 4.2 [0.00 to 9.39] | 0 [0.00 to 0.00] | 0 [0.00 to 0.00]
  Week 4 | 4.2 [0.00 to 9.39] | 3.2 [0.00 to 7.29] | 0 [0.00 to 0.00]
  Week 8: number analyzed (Participants) | 24 | 30 | 15
  Week 8 | 8.3 [1.10 to 15.56] | 6.7 [0.83 to 12.50] | 0 [0.00 to 0.00]
  Week 12: number analyzed (Participants) | 23 | 30 | 16
  Week 12 | 4.3 [0.00 to 9.80] | 6.7 [0.83 to 12.50] | 0 [0.00 to 0.00]
  Week 16: number analyzed (Participants) | 23 | 30 | 16
  Week 16 | 4.3 [0.00 to 9.80] | 3.3 [0.00 to 7.53] | 0 [0.00 to 0.00]
  Week 20: number analyzed (Participants) | 23 | 30 | 16
  Week 20 | 4.3 [0.00 to 9.80] | 6.7 [0.83 to 12.50] | 0 [0.00 to 0.00]
  Week 24: number analyzed (Participants) | 23 | 30 | 16
  Week 24 | 4.3 [0.00 to 9.80] | 6.7 [0.83 to 12.50] | 0 [0.00 to 0.00]
  Week 28: number analyzed (Participants) | 23 | 30 | 16
  Week 28 | 4.3 [0.00 to 9.80] | 3.3 [0.00 to 7.53] | 0 [0.00 to 0.00]
  Week 32: number analyzed (Participants) | 23 | 30 | 16
  Week 32 | 4.3 [0.00 to 9.80] | 3.3 [0.00 to 7.53] | 0 [0.00 to 0.00]
  Week 36: number analyzed (Participants) | 22 | 29 | 16
  Week 36 | 4.5 [0.00 to 10.24] | 3.4 [0.00 to 7.79] | 0 [0.00 to 0.00]
  Week 40: number analyzed (Participants) | 21 | 28 | 15
  Week 40 | 0 [0.00 to 0.00] | 3.6 [0.00 to 8.07] | 0 [0.00 to 0.00]
  Week 44: number analyzed (Participants) | 20 | 29 | 16
  Week 44 | 5.0 [0.00 to 11.25] | 3.4 [0.00 to 7.79] | 0 [0.00 to 0.00]
  Week 48: number analyzed (Participants) | 21 | 28 | 16
  Week 48 | 4.8 [0.00 to 10.72] | 3.6 [0.00 to 8.07] | 0 [0.00 to 0.00]
  Week 52: number analyzed (Participants) | 21 | 28 | 16
  Week 52 | 4.8 [0.00 to 10.72] | 3.6 [0.00 to 8.07] | 0 [0.00 to 0.00]
Statistical Analysis 1: Comparison: 6 mg Faricimab Q12W vs 0.5 mg Ranibizumab Q4W; Week 40: Faricimab Q12W vs. Ranibizumab Q4W; Test type: Other — The focus of this trial was estimation rather than hypothesis testing; Difference in Percentage of Participants = 0 — The difference was calculated as Faricimab Q12W arm minus Ranibizumab Q4W arm
Statistical Analysis 2: Comparison: 6 mg Faricimab Q16W vs 0.5 mg Ranibizumab Q4W; Week 40: Faricimab Q16W vs. Ranibizumab Q4W; Test type: Other — The focus of this trial was estimation rather than hypothesis testing; Difference in Percentage of Participants = 3.57, 80% CI 2-sided [-0.92 to 8.07] — The difference was calculated as Faricimab Q16W arm minus Ranibizumab Q4W arm
Statistical Analysis 3: Comparison: 6 mg Faricimab Q12W vs 0.5 mg Ranibizumab Q4W; Week 52: Faricimab Q12W vs. Ranibizumab Q4W; Test type: Other — The focus of this trial was estimation rather than hypothesis testing; Difference in Percentage of Participants = 4.76, 80% CI 2-sided [-1.19 to 10.72] — The difference was calculated as Faricimab Q12W arm minus Ranibizumab Q4W arm
Statistical Analysis 4: Comparison: 6 mg Faricimab Q16W vs 0.5 mg Ranibizumab Q4W; Week 52: Faricimab Q16W vs. Ranibizumab Q4W; Test type: Other — The focus of this trial was estimation rather than hypothesis testing; Difference in Percentage of Participants = 3.57, 80% CI 2-sided [-0.92 to 8.07] — The difference was calculated as Faricimab Q16W arm minus Ranibizumab Q4W arm

9. Secondary Outcome: Mean Change From Baseline in Central Foveal Thickness (CFT) at Specified Timepoints
Description: Central foveal thickness (CFT) was defined as the thickness from the inner limiting membrane to the retinal pigment epithelial at the horizontal slice closest to the center of the fovea, and it was measured using spectral domain optical coherence tomography (SD-OCT). The analysis was performed using a Mixed Model for Repeated Measurement (MMRM) model, which included an unstructured covariance and the categorical covariates of treatment group, visit, and visit by treatment group interaction and the continuous covariate of baseline CFT.
Time Frame: Baseline, Day 7, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: Efficacy population: participants grouped according to their assigned treatment.
Measure: Least Squares Mean (80% Confidence Interval); unit: microns (μm)
Arm/Group | 6 mg Faricimab Q12W | 6 mg Faricimab Q16W | 0.5 mg Ranibizumab Q4W
Number analyzed (Participants) | 24 | 31 | 16
microns (μm)
  Day 7 | -93.56 [-109.05 to -78.07] | -94.31 [-107.78 to -80.83] | -76.01 [-95.07 to -56.95]
  Week 4 | -132.27 [-146.13 to -118.41] | -130.11 [-142.37 to -117.85] | -122.07 [-139.47 to -104.67]
  Week 8 | -134.47 [-148.30 to -120.65] | -136.15 [-148.42 to -123.89] | -127.64 [-145.03 to -110.24]
  Week 12 | -142.26 [-157.01 to -127.52] | -139.63 [-152.66 to -126.59] | -126.63 [-145.03 to -108.24]
  Week 16 | -134.94 [-150.26 to -119.63] | -137.81 [-151.37 to -124.25] | -120.48 [-139.55 to -101.40]
  Week 20 | -125.05 [-143.75 to -106.35] | -125.35 [-141.86 to -108.84] | -120.70 [-143.69 to -97.70]
  Week 24 | -121.13 [-140.94 to -101.31] | -108.66 [-126.14 to -91.17] | -131.29 [-155.62 to -106.96]
  Week 28 | -131.58 [-148.18 to -114.99] | -116.76 [-131.41 to -102.12] | -130.29 [-150.80 to -109.78]
  Week 32 | -127.85 [-149.31 to -106.38] | -123.44 [-142.37 to -104.51] | -134.29 [-160.61 to -107.97]
  Week 36 | -114.27 [-134.82 to -93.71] | -114.97 [-133.02 to -96.92] | -149.26 [-174.17 to -124.35]
  Week 40 | -137.54 [-156.68 to -118.40] | -123.31 [-140.20 to -106.42] | -137.99 [-161.27 to -114.71]
  Week 44 | -135.30 [-154.78 to -115.82] | -110.26 [-127.23 to -93.30] | -135.70 [-159.16 to -112.23]
  Week 48 | -125.93 [-145.69 to -106.17] | -121.67 [-139.07 to -104.26] | -130.76 [-154.93 to -106.58]
  Week 52 | -140.95 [-157.06 to -124.85] | -134.99 [-149.21 to -120.76] | -136.10 [-155.98 to -116.23]
Statistical Analysis 1: Comparison: 6 mg Faricimab Q12W vs 0.5 mg Ranibizumab Q4W; Week 40: Faricimab Q12W vs. Ranibizumab Q4W; Test type: Other — The focus of this trial was estimation rather than hypothesis testing; Mean Difference (Net) = 0.45, 80% CI 2-sided [-29.81 to 30.71] — The difference was calculated as Faricimab Q12W arm minus Ranibizumab Q4W arm
Statistical Analysis 2: Comparison: 6 mg Faricimab Q16W vs 0.5 mg Ranibizumab Q4W; Week 40: Faricimab Q16W vs. Ranibizumab Q4W; Test type: Other — The focus of this trial was estimation rather than hypothesis testing; Mean Difference (Net) = 14.68, 80% CI 2-sided [-14.29 to 43.65] — The difference was calculated as Faricimab Q16W arm minus Ranibizumab Q4W arm
Statistical Analysis 3: Comparison: 6 mg Faricimab Q12W vs 0.5 mg Ranibizumab Q4W; Week 52: Faricimab Q12W vs. Ranibizumab Q4W; Test type: Other — The focus of this trial was estimation rather than hypothesis testing; Mean Difference (Net) = -4.85, 80% CI 2-sided [-30.57 to 20.87] — The difference was calculated as Faricimab Q12W arm minus Ranibizumab Q4W arm
Statistical Analysis 4: Comparison: 6 mg Faricimab Q16W vs 0.5 mg Ranibizumab Q4W; Week 52: Faricimab Q16W vs. Ranibizumab Q4W; Test type: Other — The focus of this trial was estimation rather than hypothesis testing; Mean Difference (Net) = 1.12, 80% CI 2-sided [-23.57 to 25.80] — The difference was calculated as Faricimab Q16W arm minus Ranibizumab Q4W arm

10. Secondary Outcome: Mean Change From Baseline in Central Subfield Thickness (CST) at Specified Timepoints
Description: Central subfield thickness (CST) was defined as the mean thickness from the inner limiting membrane to the retinal pigment epithelial over the 1 millimetre (mm) central subfield, and it was measured using spectral domain optical coherence tomography (SD-OCT). The analysis was performed using a Mixed Model for Repeated Measurement (MMRM) model, which included an unstructured covariance and the categorical covariates of treatment group, visit, and visit by treatment group interaction and the continuous covariate of baseline CST.
Time Frame: Baseline, Day 7, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: Efficacy population: participants grouped according to their assigned treatment.
Measure: Least Squares Mean (80% Confidence Interval); unit: microns (μm)
Arm/Group | 6 mg Faricimab Q12W | 6 mg Faricimab Q16W | 0.5 mg Ranibizumab Q4W
Number analyzed (Participants) | 24 | 31 | 16
microns (μm)
  Day 7 | -88.87 [-100.40 to -77.34] | -84.23 [-94.35 to -74.11] | -80.08 [-94.15 to -66.01]
  Week 4 | -127.20 [-139.69 to -114.72] | -123.10 [-134.18 to -112.02] | -111.58 [-126.99 to -96.17]
  Week 8 | -132.03 [-145.40 to -118.67] | -131.25 [-143.13 to -119.37] | -117.04 [-133.54 to -100.53]
  Week 12 | -134.70 [-148.96 to -120.44] | -132.87 [-145.53 to -120.20] | -122.39 [-139.93 to -104.85]
  Week 16 | -132.96 [-147.69 to -118.23] | -132.50 [-145.58 to -119.42] | -122.70 [-140.81 to -104.60]
  Week 20 | -114.97 [-131.83 to -98.12] | -118.89 [-133.77 to -104.00] | -120.77 [-141.28 to -100.25]
  Week 24 | -101.62 [-119.69 to -83.54] | -99.35 [-115.29 to -83.42] | -121.33 [-143.26 to -99.40]
  Week 28 | -129.68 [-144.40 to -114.95] | -109.89 [-122.91 to -96.87] | -127.95 [-145.93 to -109.98]
  Week 32 | -121.10 [-139.50 to -102.71] | -116.35 [-132.57 to -100.14] | -127.20 [-149.56 to -104.85]
  Week 36 | -101.98 [-121.60 to -82.36] | -102.69 [-119.96 to -85.42] | -118.89 [-142.63 to -95.15]
  Week 40 | -138.55 [-154.04 to -123.05] | -121.34 [-135.07 to -107.62] | -126.32 [-145.20 to -107.44]
  Week 44 | -130.50 [-146.19 to -114.81] | -103.31 [-117.04 to -89.57] | -124.89 [-143.71 to -106.08]
  Week 48 | -126.45 [-145.58 to -107.33] | -102.30 [-119.14 to -85.47] | -123.89 [-147.01 to -100.77]
  Week 52 | -138.53 [-152.42 to -124.65] | -122.53 [-134.81 to -110.25] | -129.89 [-146.74 to -113.04]
Statistical Analysis 1: Comparison: 6 mg Faricimab Q12W vs 0.5 mg Ranibizumab Q4W; Week 40: Faricimab Q12W vs. Ranibizumab Q4W; Test type: Other — The focus of this trial was estimation rather than hypothesis testing; Mean Difference (Net) = -12.23, 80% CI 2-sided [-36.60 to 12.15] — The difference was calculated as Faricimab Q12W arm minus Ranibizumab Q4W arm
Statistical Analysis 2: Comparison: 6 mg Faricimab Q16W vs 0.5 mg Ranibizumab Q4W; Week 40: Faricimab Q16W vs. Ranibizumab Q4W; Test type: Other — The focus of this trial was estimation rather than hypothesis testing; Mean Difference (Net) = 4.98, 80% CI 2-sided [-18.50 to 28.45] — The difference was calculated as Faricimab Q16W arm minus Ranibizumab Q4W arm
Statistical Analysis 3: Comparison: 6 mg Faricimab Q12W vs 0.5 mg Ranibizumab Q4W; Week 52: Faricimab Q12W vs. Ranibizumab Q4W; Test type: Other — The focus of this trial was estimation rather than hypothesis testing; Mean Difference (Net) = -8.64, 80% CI 2-sided [-30.42 to 13.14] — The difference was calculated as Faricimab Q12W arm minus Ranibizumab Q4W arm
Statistical Analysis 4: Comparison: 6 mg Faricimab Q16W vs 0.5 mg Ranibizumab Q4W; Week 52: Faricimab Q16W vs. Ranibizumab Q4W; Test type: Other — The focus of this trial was estimation rather than hypothesis testing; Mean Difference (Net) = 7.36, 80% CI 2-sided [-13.65 to 28.37] — The difference was calculated as Faricimab Q16W arm minus Ranibizumab Q4W arm

11. Secondary Outcome: Percentage of Participants With No Intraretinal Fluid at Specified Timepoints
Description: The absence of intraretinal fluid, subretinal fluid, cysts, or pigment epithelial detachment, as per the study's dry retina definition, were evaluated as individual dry retina outcomes. Intraretinal fluid was defined as the presence of fluid within the retina. All parameters were measured using spectral domain optical coherence tomography (SD-OCT). Anatomic outcome measures were based on results from a central reading center. This analysis was performed on observed data. The 80% confidence intervals were calculated using the Wald method.
Time Frame: Baseline, Day 7, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: as for outcome 3
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | 6 mg Faricimab Q12W | 6 mg Faricimab Q16W | 0.5 mg Ranibizumab Q4W
Number analyzed (Participants) | 24 | 31 | 16
Percentage of participants
  Baseline | 4.2 [0.00 to 9.39] | 29.0 [18.58 to 39.48] | 18.8 [6.24 to 31.26]
  Day 7: number analyzed (Participants) | 23 | 31 | 16
  Day 7 | 21.7 [10.72 to 32.76] | 38.7 [27.50 to 49.92] | 25.0 [11.13 to 38.87]
  Week 4 | 29.2 [17.28 to 41.06] | 48.4 [36.88 to 59.89] | 50.0 [33.98 to 66.02]
  Week 8: number analyzed (Participants) | 24 | 30 | 15
  Week 8 | 33.3 [21.00 to 45.67] | 46.7 [34.99 to 58.34] | 26.7 [12.03 to 41.30]
  Week 12: number analyzed (Participants) | 23 | 30 | 16
  Week 12 | 39.1 [26.09 to 52.17] | 43.3 [31.74 to 54.93] | 37.5 [21.99 to 53.01]
  Week 16: number analyzed (Participants) | 23 | 30 | 16
  Week 16 | 47.8 [34.48 to 61.17] | 50.0 [38.30 to 61.70] | 37.5 [21.99 to 53.01]
  Week 20: number analyzed (Participants) | 23 | 30 | 16
  Week 20 | 43.5 [30.23 to 56.73] | 53.3 [41.66 to 65.01] | 18.8 [6.24 to 31.26]
  Week 24: number analyzed (Participants) | 23 | 30 | 16
  Week 24 | 30.4 [18.14 to 42.73] | 50.0 [38.30 to 61.70] | 31.3 [16.40 to 46.10]
  Week 28: number analyzed (Participants) | 23 | 30 | 16
  Week 28 | 26.1 [14.35 to 37.82] | 53.3 [41.66 to 65.01] | 31.3 [16.40 to 46.10]
  Week 32: number analyzed (Participants) | 23 | 30 | 16
  Week 32 | 26.1 [14.35 to 37.82] | 50.0 [38.30 to 61.70] | 31.3 [16.40 to 46.10]
  Week 36: number analyzed (Participants) | 22 | 29 | 16
  Week 36 | 31.8 [19.09 to 44.54] | 44.8 [32.99 to 56.66] | 37.5 [21.99 to 53.01]
  Week 40: number analyzed (Participants) | 21 | 28 | 15
  Week 40 | 38.1 [24.51 to 51.68] | 57.1 [45.16 to 69.13] | 33.3 [17.73 to 48.93]
  Week 44: number analyzed (Participants) | 20 | 29 | 16
  Week 44 | 55.0 [40.74 to 69.26] | 48.3 [36.38 to 60.17] | 43.8 [27.86 to 59.64]
  Week 48: number analyzed (Participants) | 21 | 28 | 16
  Week 48 | 38.1 [24.51 to 51.68] | 53.6 [41.49 to 65.65] | 62.5 [46.99 to 78.01]
  Week 52: number analyzed (Participants) | 21 | 28 | 16
  Week 52 | 38.1 [24.51 to 51.68] | 35.7 [24.11 to 47.32] | 62.5 [46.99 to 78.01]

12. Secondary Outcome: Percentage of Participants With No Subretinal Fluid at Specified Timepoints
Description: The absence of intraretinal fluid, subretinal fluid, cysts, or pigment epithelial detachment, as per the study's dry retina definition, were evaluated as individual dry retina outcomes. Subretinal fluid was defined as the presence of fluid between the retina and the retinal pigment epithelium. All parameters were measured using spectral domain optical coherence tomography (SD-OCT). Anatomic outcome measures were based on results from a central reading center. This analysis was performed on observed data. The 80% confidence intervals were calculated using the Wald method.
Time Frame: Baseline, Day 7, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: as for outcome 3
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | 6 mg Faricimab Q12W | 6 mg Faricimab Q16W | 0.5 mg Ranibizumab Q4W
Number analyzed (Participants) | 24 | 31 | 16
Percentage of participants
  Baseline | 20.8 [10.21 to 31.46] | 12.9 [5.19 to 20.62] | 25.0 [11.13 to 38.87]
  Day 7: number analyzed (Participants) | 23 | 31 | 16
  Day 7 | 39.1 [26.09 to 52.17] | 29.0 [18.58 to 39.48] | 31.3 [16.40 to 46.10]
  Week 4 | 70.8 [58.94 to 82.72] | 77.4 [67.80 to 87.04] | 62.5 [46.99 to 78.01]
  Week 8: number analyzed (Participants) | 24 | 30 | 15
  Week 8 | 83.3 [73.58 to 93.08] | 86.7 [78.71 to 94.62] | 80.0 [66.76 to 93.24]
  Week 12: number analyzed (Participants) | 23 | 30 | 16
  Week 12 | 91.3 [83.77 to 98.83] | 90.0 [82.98 to 97.02] | 75.0 [61.13 to 88.87]
  Week 16: number analyzed (Participants) | 23 | 30 | 16
  Week 16 | 87.0 [77.96 to 95.96] | 96.7 [92.47 to 100.00] | 75.0 [61.13 to 88.87]
  Week 20: number analyzed (Participants) | 23 | 30 | 16
  Week 20 | 69.6 [57.27 to 81.86] | 70.0 [59.28 to 80.72] | 87.5 [76.90 to 98.10]
  Week 24: number analyzed (Participants) | 23 | 30 | 16
  Week 24 | 65.2 [52.49 to 77.94] | 66.7 [55.64 to 77.70] | 75.0 [61.13 to 88.87]
  Week 28: number analyzed (Participants) | 23 | 30 | 16
  Week 28 | 91.3 [83.77 to 98.83] | 70.0 [59.28 to 80.72] | 75.0 [61.13 to 88.87]
  Week 32: number analyzed (Participants) | 23 | 30 | 16
  Week 32 | 69.6 [57.27 to 81.86] | 80.0 [70.64 to 89.36] | 68.8 [53.90 to 83.60]
  Week 36: number analyzed (Participants) | 22 | 29 | 16
  Week 36 | 68.2 [55.46 to 80.91] | 72.4 [61.78 to 83.05] | 81.3 [68.74 to 93.76]
  Week 40: number analyzed (Participants) | 21 | 28 | 15
  Week 40 | 81.0 [69.97 to 91.93] | 89.3 [81.79 to 96.78] | 86.7 [75.42 to 97.91]
  Week 44: number analyzed (Participants) | 20 | 29 | 16
  Week 44 | 80.0 [68.54 to 91.46] | 75.9 [65.68 to 86.05] | 81.3 [68.74 to 93.76]
  Week 48: number analyzed (Participants) | 21 | 28 | 16
  Week 48 | 71.4 [58.79 to 84.06] | 64.3 [52.68 to 75.89] | 87.5 [76.90 to 98.10]
  Week 52: number analyzed (Participants) | 21 | 28 | 16
  Week 52 | 81.0 [69.97 to 91.93] | 89.3 [81.79 to 96.78] | 87.5 [76.90 to 98.10]

13. Secondary Outcome: Percentage of Participants With No Cysts at Specified Timepoints
Description: The absence of intraretinal fluid, subretinal fluid, cysts, or pigment epithelial detachment, as per the study's dry retina definition, were evaluated as individual dry retina outcomes. Cysts were defined as the presence of cystoid space (fluid) in the retina. All parameters were measured using spectral domain optical coherence tomography (SD-OCT). Anatomic outcome measures were based on results from a central reading center. This analysis was performed on observed data. The 80% confidence intervals were calculated using the Wald method.
Time Frame: Baseline, Day 7, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: as for outcome 3
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | 6 mg Faricimab Q12W | 6 mg Faricimab Q16W | 0.5 mg Ranibizumab Q4W
Number analyzed (Participants) | 24 | 31 | 16
Percentage of participants
  Baseline | 33.3 [21.00 to 45.67] | 48.4 [36.88 to 59.89] | 37.5 [21.99 to 53.01]
  Day 7: number analyzed (Participants) | 23 | 31 | 16
  Day 7 | 65.2 [52.49 to 77.94] | 83.9 [75.41 to 92.34] | 75.0 [61.13 to 88.87]
  Week 4 | 87.5 [78.85 to 96.15] | 87.1 [79.38 to 94.81] | 87.5 [76.90 to 98.10]
  Week 8: number analyzed (Participants) | 24 | 30 | 15
  Week 8 | 83.3 [73.58 to 93.08] | 83.3 [74.61 to 92.05] | 86.7 [75.42 to 97.91]
  Week 12: number analyzed (Participants) | 23 | 30 | 16
  Week 12 | 91.3 [83.77 to 98.83] | 83.3 [74.61 to 92.05] | 68.8 [53.90 to 83.60]
  Week 16: number analyzed (Participants) | 23 | 30 | 16
  Week 16 | 91.3 [83.77 to 98.83] | 83.3 [74.61 to 92.05] | 75.0 [61.13 to 88.87]
  Week 20: number analyzed (Participants) | 23 | 30 | 16
  Week 20 | 91.3 [83.77 to 98.83] | 80.0 [70.64 to 89.36] | 68.8 [53.90 to 83.60]
  Week 24: number analyzed (Participants) | 23 | 30 | 16
  Week 24 | 73.9 [62.18 to 85.65] | 76.7 [66.77 to 86.56] | 68.8 [53.90 to 83.60]
  Week 28: number analyzed (Participants) | 23 | 30 | 16
  Week 28 | 95.7 [90.20 to 100.00] | 70.0 [59.28 to 80.72] | 68.8 [53.90 to 83.60]
  Week 32: number analyzed (Participants) | 23 | 30 | 16
  Week 32 | 82.6 [72.48 to 92.74] | 76.7 [66.77 to 86.56] | 75.0 [61.13 to 88.87]
  Week 36: number analyzed (Participants) | 22 | 29 | 16
  Week 36 | 77.3 [65.82 to 88.72] | 79.3 [69.67 to 88.95] | 68.8 [53.90 to 83.60]
  Week 40: number analyzed (Participants) | 21 | 28 | 15
  Week 40 | 85.7 [75.93 to 95.50] | 78.6 [68.63 to 88.51] | 80.0 [66.76 to 93.24]
  Week 44: number analyzed (Participants) | 20 | 29 | 16
  Week 44 | 100.0 [100.00 to 100.00] | 72.4 [61.78 to 83.05] | 87.5 [76.90 to 98.10]
  Week 48: number analyzed (Participants) | 21 | 28 | 16
  Week 48 | 95.2 [89.28 to 100.00] | 85.7 [77.24 to 94.19] | 87.5 [76.90 to 98.10]
  Week 52: number analyzed (Participants) | 21 | 28 | 16
  Week 52 | 100.0 [100.00 to 100.00] | 78.6 [68.63 to 88.51] | 87.5 [76.90 to 98.10]

14. Secondary Outcome: Percentage of Participants With No Pigment Epithelial Detachment at Specified Timepoints
Description: The absence of intraretinal fluid, subretinal fluid, cysts, or pigment epithelial detachment, as per the study's dry retina definition, were evaluated as individual dry retina outcomes. Pigment epithelial detachment was defined as the presence of a detachment of the pigment epithelium from the Bruch's membrane. All parameters were measured using spectral domain optical coherence tomography (SD-OCT). Anatomic outcome measures were based on results from a central reading center. This analysis was performed on observed data. The 80% confidence intervals were calculated using the Wald method.
Time Frame: Baseline, Day 7, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: as for outcome 3
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | 6 mg Faricimab Q12W | 6 mg Faricimab Q16W | 0.5 mg Ranibizumab Q4W
Number analyzed (Participants) | 24 | 31 | 16
Percentage of participants
  Baseline | 8.3 [1.10 to 15.56] | 29.0 [18.58 to 39.48] | 12.5 [1.90 to 23.10]
  Day 7: number analyzed (Participants) | 23 | 31 | 16
  Day 7 | 13.0 [4.04 to 22.04] | 29.0 [18.58 to 39.48] | 12.5 [1.90 to 23.10]
  Week 4 | 8.3 [1.10 to 15.56] | 22.6 [12.96 to 32.20] | 12.5 [1.90 to 23.10]
  Week 8: number analyzed (Participants) | 24 | 30 | 15
  Week 8 | 8.3 [1.10 to 15.56] | 23.3 [13.44 to 33.23] | 13.3 [2.09 to 24.58]
  Week 12: number analyzed (Participants) | 23 | 30 | 16
  Week 12 | 8.7 [1.17 to 16.23] | 26.7 [16.32 to 37.01] | 12.5 [1.90 to 23.10]
  Week 16: number analyzed (Participants) | 23 | 30 | 16
  Week 16 | 8.7 [1.17 to 16.23] | 23.3 [13.44 to 33.23] | 12.5 [1.90 to 23.10]
  Week 20: number analyzed (Participants) | 23 | 30 | 16
  Week 20 | 13.0 [4.04 to 22.04] | 23.3 [13.44 to 33.23] | 12.5 [1.90 to 23.10]
  Week 24: number analyzed (Participants) | 23 | 30 | 16
  Week 24 | 13.0 [4.04 to 22.04] | 23.3 [13.44 to 33.23] | 12.5 [1.90 to 23.10]
  Week 28: number analyzed (Participants) | 23 | 30 | 16
  Week 28 | 13.0 [4.04 to 22.04] | 20.0 [10.64 to 29.36] | 12.5 [1.90 to 23.10]
  Week 32: number analyzed (Participants) | 23 | 30 | 16
  Week 32 | 13.0 [4.04 to 22.04] | 23.3 [13.44 to 33.23] | 12.5 [1.90 to 23.10]
  Week 36: number analyzed (Participants) | 22 | 29 | 16
  Week 36 | 4.5 [0.00 to 10.24] | 20.7 [11.05 to 30.33] | 12.5 [1.90 to 23.10]
  Week 40: number analyzed (Participants) | 21 | 28 | 15
  Week 40 | 4.8 [0.00 to 10.72] | 21.4 [11.49 to 31.37] | 13.3 [2.09 to 24.58]
  Week 44: number analyzed (Participants) | 20 | 29 | 16
  Week 44 | 5.0 [0.00 to 11.25] | 17.2 [8.25 to 26.23] | 12.5 [1.90 to 23.10]
  Week 48: number analyzed (Participants) | 21 | 28 | 16
  Week 48 | 9.5 [1.31 to 17.73] | 17.9 [8.58 to 27.13] | 12.5 [1.90 to 23.10]
  Week 52: number analyzed (Participants) | 21 | 28 | 16
  Week 52 | 14.3 [4.50 to 24.07] | 14.3 [5.81 to 22.76] | 12.5 [1.90 to 23.10]

15. Secondary Outcome: Mean Baseline Value and Mean Change From Baseline of Total Area of Choroidal Neovascularization (CNV) at Week 40 and Week 52
Description: The total area of choroidal neovascularization (CNV) was evaluated by a central reading center using fundus fluorescein angiography (FFA).
Time Frame: Baseline, Week 40, Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimetres squared (mm^2)
Arm/Group | 6 mg Faricimab Q12W | 6 mg Faricimab Q16W | 0.5 mg Ranibizumab Q4W
Number analyzed (Participants) | 24 | 31 | 16
millimetres squared (mm^2)
  Baseline (BL): Absolute Value | 7.1 (3.9) | 5.9 (3.8) | 7.3 (2.9)
  Change from BL at Week 40: number analyzed (Participants) | 19 | 26 | 14
  Change from BL at Week 40 | -4.7 (4.3) | -3.9 (3.7) | -4.6 (3.5)
  Change from BL at Week 52: number analyzed (Participants) | 19 | 28 | 16
  Change from BL at Week 52 | -5.4 (4.0) | -4.2 (3.4) | -4.5 (3.2)

16. Secondary Outcome: Mean Baseline Value and Mean Change From Baseline of Total Area of CNV Component at Week 40 and Week 52
Description: The total area of choroidal neovascularization (CNV) component (i.e., total area of CNV membrane) was evaluated by a central reading center using fundus fluorescein angiography (FFA).
Time Frame: Baseline, Week 40, Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimetres squared (mm^2)
Arm/Group | 6 mg Faricimab Q12W | 6 mg Faricimab Q16W | 0.5 mg Ranibizumab Q4W
Number analyzed (Participants) | 24 | 31 | 16
millimetres squared (mm^2)
  Baseline (BL): Absolute Value | 7.0 (3.8) | 5.8 (3.6) | 7.1 (3.0)
  Change from BL at Week 40: number analyzed (Participants) | 19 | 26 | 14
  Change from BL at Week 40 | -5.0 (4.2) | -4.0 (4.0) | -4.7 (3.4)
  Change from BL at Week 52: number analyzed (Participants) | 19 | 28 | 16
  Change from BL at Week 52 | -5.6 (4.0) | -4.3 (3.7) | -4.8 (3.2)

17. Secondary Outcome: Mean Baseline Value and Mean Change From Baseline of Total Area of Leakage at Week 40 and Week 52
Description: The total area of leakage was evaluated by a central reading center using fundus fluorescein angiography (FFA).
Time Frame: Baseline, Week 40, Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimetres squared (mm^2)
Arm/Group | 6 mg Faricimab Q12W | 6 mg Faricimab Q16W | 0.5 mg Ranibizumab Q4W
Number analyzed (Participants) | 24 | 31 | 16
millimetres squared (mm^2)
  Baseline (BL): Absolute Value | 7.0 (3.8) | 6.1 (3.4) | 7.6 (2.9)
  Change from BL at Week 40: number analyzed (Participants) | 19 | 26 | 14
  Change from BL at Week 40 | -5.0 (4.2) | -4.3 (3.9) | -5.3 (3.7)
  Change from BL at Week 52: number analyzed (Participants) | 19 | 28 | 16
  Change from BL at Week 52 | -5.6 (4.0) | -4.6 (3.5) | -5.3 (3.5)

18. Secondary Outcome: Change From Baseline in the Number of Participants With Anti-Drug Antibodies (ADA) to Faricimab at Anytime Post-Baseline
Description: Blood samples were obtained for measurement of anti-drug antibodies (ADAs) to faricimab by a validated enzyme-linked immunosorbent assay (ELISA).
Time Frame: Predose at Baseline (Day 1), Weeks 16, 24, 28, 44, and 52
Population: Safety Population: participants who received at least one dose of study treatment, grouped according to treatment received. The analysis only included participants who received treatment with faricimab (i.e., 0.5 mg Ranibizumab Q4W arm was excluded) and had evaluable samples at baseline and/or any post-baseline timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | 6 mg Faricimab Q12W | 6 mg Faricimab Q16W
Number analyzed (Participants) | 24 | 31
Participants
  ADA Negative to ADA Negative | 21 | 25
  ADA Negative to ADA Positive | 1 | 4
  Missing to ADA Negative | 0 | 1
  Missing to ADA Positive | 1 | 0
  No Post-Baseline ADA Assessment | 1 | 1

19. Secondary Outcome: Safety Summary: Number and Percentage of Participants With at Least One Adverse Event
Description: This safety summary reports the number and percentage of participants who experienced at least one adverse event (AE) during the study. The investigator independently assessed the seriousness and severity for each AE. Severity was graded according to the following grading scale: Mild = Discomfort noticed, but no disruption of normal daily activity; Moderate = Discomfort sufficient to reduce or affect normal daily activity; Severe = Incapacitating with inability to work or to perform normal daily activity. Severity and seriousness are not synonymous; regardless of severity, some AEs may have also met seriousness criteria.
Time Frame: From Baseline until 28 days after the last dose of study drug (up to 52 weeks)
Population: Safety Population: participants who received at least one dose of the study treatment, grouped according to treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | 6 mg Faricimab Q12W | 6 mg Faricimab Q16W | 0.5 mg Ranibizumab Q4W
Number analyzed (Participants) | 24 | 31 | 16
Participants
  Any Adverse Event (AE) | 18 | 23 | 13
  Serious AE (SAE) | 4 | 3 | 0
  SAE Leading to Withdrawal from Treatment | 0 | 0 | 0
  SAE Leading to Dose Modification/Interruption | 1 | 0 | 0
  Serious Ocular AE | 0 | 0 | 0
  Serious Non-Ocular AE | 4 | 3 | 0
  AE Leading to Withdrawal from Treatment | 0 | 0 | 0
  AE Leading to Dose Modification/Interruption | 2 | 0 | 0
  Ocular AE in the Study Eye | 9 | 11 | 8
  Ocular AE in the Fellow Eye | 6 | 5 | 6
  Non-Ocular AE | 14 | 20 | 9

ADVERSE EVENTS:
Time Frame: From Baseline until 28 days after the last dose of study drug (up to 52 weeks)
Arm/Group | 6 mg Faricimab Q12W | 6 mg Faricimab Q16W | 0.5 mg Ranibizumab Q4W
All-Cause Mortality (participants affected / at risk) | 1/24 | 2/31 | 0/16
Serious Adverse Events (participants affected / at risk) | 4/24 | 3/31 | 0/16
Other Adverse Events (participants affected / at risk) | 18/24 | 22/31 | 13/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 6 mg Faricimab Q12W (N=24) | 6 mg Faricimab Q16W (N=31) | 0.5 mg Ranibizumab Q4W (N=16)
Acute left ventricular failure (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 6 mg Faricimab Q12W (N=24) | 6 mg Faricimab Q16W (N=31) | 0.5 mg Ranibizumab Q4W (N=16)
Conjunctival haemorrhage (Eye disorders) | 5 | 4 | 4
Neovascular age-related macular degeneration (Eye disorders) | 3 | 0 | 2
Eye pain (Eye disorders) | 2 | 0 | 2
Retinal haemorrhage (Eye disorders) | 2 | 0 | 2
Cataract (Eye disorders) | 2 | 1 | 0
Choroidal neovascularisation (Eye disorders) | 1 | 0 | 1
Dry eye (Eye disorders) | 0 | 1 | 1
Maculopathy (Eye disorders) | 0 | 2 | 0
Ocular discomfort (Eye disorders) | 0 | 1 | 1
Vitreous detachment (Eye disorders) | 1 | 0 | 1
Vitreous floaters (Eye disorders) | 1 | 0 | 1
Eye haemorrhage (Eye disorders) | 0 | 0 | 1
Macular oedema (Eye disorders) | 0 | 0 | 1
Ocular hypertension (Eye disorders) | 0 | 0 | 1
Optic disc haemorrhage (Eye disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 4 | 2 | 1
Urinary tract infection (Infections and infestations) | 1 | 2 | 1
Influenza (Infections and infestations) | 1 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 1
Vaginal infection (Infections and infestations) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 5 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 2 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Eye contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 1 | 1
Cyst (General disorders) | 0 | 0 | 1
Biopsy palate (Investigations) | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 2 | 0
Hypothyroidism (Endocrine disorders) | 0 | 2 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Anterior chamber flare (Eye disorders) | 1 | 0 | 0
Chalazion (Eye disorders) | 1 | 0 | 0
Eye irritation (Eye disorders) | 1 | 0 | 0
Eye pruritus (Eye disorders) | 1 | 0 | 0
Foreign body sensation in eyes (Eye disorders) | 0 | 1 | 0
Iritis (Eye disorders) | 0 | 1 | 0
Subretinal fibrosis (Eye disorders) | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 1 | 0 | 0
Punctate keratitis (Eye disorders) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0
Catheter site infection (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Joint abscess (Infections and infestations) | 0 | 1 | 0
Mycobacterium avium complex infection (Infections and infestations) | 1 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0
Urethritis (Infections and infestations) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0
Inflammatory pain (General disorders) | 0 | 1 | 0
Blood sodium decreased (Investigations) | 0 | 1 | 0
Catheterisation cardiac (Investigations) | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Cerebral small vessel ischaemic disease (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Bladder pain (Renal and urinary disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Chorioretinal atrophy (Eye disorders) | 1 | 0 | 0
Macular fibrosis (Eye disorders) | 0 | 1 | 0
Retinal drusen (Eye disorders) | 0 | 1 | 0
Vitreous disorder (Eye disorders) | 0 | 1 | 0
Eye naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Aneurysm (Vascular disorders) | 0 | 1 | 0
Intraocular pressure increased (Investigations) | 0 | 0 | 1
Ophthalmological examination abnormal (Investigations) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Interpretability of the imaging endpoints is limited by the relatively small sample size of the study and imbalances between the arms at baseline. Formal comparisons could not be performed across the treatment arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-14): https://cdn.clinicaltrials.gov/large-docs/80/NCT03038880/Prot_SAP_000.pdf